CLINICAL TRIAL: NCT01862588
Title: Clinical Study of Renal Resistive Index and Hemodynamic Parameters Changes Caused by Fluid Resuscitation to Predict the Occurrence of Acute Kidney Injury in Septic Shock Patients
Brief Title: Renal Resistive Index and Cardiac Output Changes During Resuscitation Predict the Occurrence of Acute Kidney Injury in Septic Shock Patients
Acronym: CORRI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Xiaohua Qiu, physician, Zhongda Hospital
Other Study IDs: 201314159
Record Dates: First submitted 2013-05-13; First posted 2013-05-24 (Estimated); Last update posted 2014-01-15 (Estimated); Status verified 2014-01

CONDITIONS: Critically Ill; Acute Kidney Injury; Septic Shock
Keywords: septic shock; acute kidney injury; renal resistive index
MeSH Terms: conditions — Critical Illness; Acute Kidney Injury; Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — For every enrolled patient,we will collect 5ml blood plasma for renal function examination, and this point will fully informed and approved by the Ethic Committee.
Oversight: Data Monitoring Committee: No

SUMMARY:
Record the renal resistive index and hemodynamic parameters ( record the cardiac output and stroke volume if the patient's next to kin agree to undertake a PiCCO monitoring ) before and after resuscitation for severe sepsis or septic shock patients, to determine whether the changes of resistive index or hemodynamic parameters, especially the cardiac output can be a better parameter to predict AKI

DETAILED DESCRIPTION:
* Purpose: To examine whether the resuscitation-induced changes of renal resistive index or hemodynamic parameters has the superiority as a valid tool to evaluate the renal perfusion improvement and whether the changes can better predict AKI occurrence in severe sepsis or septic shock patients.
* Methods: Measure the renal resistive index and take record of hemodynamic parameters (use a PiCCO monitoring to measure cardiac output if the patient's next to kin agree to undertake such a catheter ) before and after successful resuscitation for severe sepsis or septic shock patients, followup to determine the occurrence of AKI and mortality.
* Hypothesis: The changes of resistive index or cardiac output during shock resuscitation may be a better parameter to evaluate renal perfusion and predict AKI, and may have a better value to guide renal protective therapy in septic shock.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years, Sex unlimited
* Arriving ICU in 6 hours and diagnosed with severe sepsis or septic shock
* Physician in charge decide that an aggressive fluid resuscitation was in order

Exclusion Criteria:

* Pregnancy, Age <18 years
* Ongoing recovery from AKI
* Known end-stage renal disease or chronic kidney disease(glomerular filtration rate <30mL/min/1.73m2)
* Known other causes of shock morbidly
* conditions known to modify RRI, such as renal-artery stenosis, intra-abdominal hypertension(>35cmH2O)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critical ill patients diagnosed with septic shock who required a fluid resuscitation.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-01 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
7 days AKI occurrence | 7 days
  Follow up to determine the occurrence of AKI in 7 days after inclusion.

SECONDARY OUTCOMES:
eGFR | until 6 hours after enrollment
  eGFR when enrolled and 6 hours after enrollment.The 2012 SSC guideline for severe sepsis and septic shock recommend to achieve some six-hour resuscitation goals.So we collect 5ml blood and 2 hrs urine when enrolled(at this time, initiate large amount of fluid resuscitation,which is so called "before resuscitation"). At 6hrs after enrolled,collect another 5ml blood and 2 hrs urine.Glomerular filtration rate (GFR) describes the flow rate of filtered fluid through the kidney. eGFR is Creatinine-based approximations of GFR. We project to use the "Urine Creatinine concentration×Urine Flow Rate/Plasma Creatinine Concentration" formula to calculate the eGFR (collected two hours urine, and examine the plasma and urine creatinine in the middle of the two hours). The lowest plasma creatinine value in the 3 months preceding inclusion was taken as the baseline value, therefore use the value to calculate baseline eGFR by CKD-EPI formula.

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Zhongda Hospital of Southeast University, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Luo JC, Qiu XH, Pan C, Xie JF, Yu T, Liu L, Yang Y, Qiu HB. Increased cardiac index attenuates septic acute kidney injury: a prospective observational study. BMC Anesthesiol. 2015 Mar 1;15:22. doi: 10.1186/s12871-015-0005-0. eCollection 2015. PMID 25745357